CLINICAL TRIAL: NCT03759678
Title: Effects of N-Acetyl-L-Leucine on Ataxia-Telangiectasia (A-T): A Multinational, Multicenter, Open-label, Rater-blinded Phase II Study
Brief Title: N-Acetyl-L-Leucine for Ataxia-Telangiectasia (A-T)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IntraBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IB1001-203
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Ataxia Telangiectasia; Louis Bar Syndrome
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — IB1001; acetylleucine

STUDY DESIGN:
Intervention Model Description: Patients will be assessed during three study phases: a baseline period (with or without a study run-in), a treatment period, and a washout period.
Who Masked: Outcomes Assessor
Masking Description: The primary evaluation of the Clinical Impression of Change in Severity (CI-CS; Primary Endpoint) will be performed by two independent neurologists whose assessments are based on videos of patient's performance on either the 9 Hole Peg Test of the Dominant Hand (9HPT-D) or the 8 Meter Walk Test (8MWT) taken at each visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with IB1001 (Experimental): 6-weeks treatment with IB1001 administered orally.
  Patients ≥13 years old will receive a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old will receive weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg will take 2 g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg will take 3 g per day: 1 g in the morning, 1 g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg will take 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  After the 6-week treatment period, patients will enter a 6-week post-treatment washout period.
  Interventions: Drug: IB1001
- Post-Treatment Washout (No Intervention): After the 6-week treatment period, patients will enter a 6-week post-treatment washout period.

INTERVENTIONS:
Drug: IB1001 — IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  Other Names: N-Acetyl-L-Leucine
  Arms: Treatment with IB1001

SUMMARY:
This is a multinational, multicenter, open-label, rater-blinded prospective Phase II study which will assess the safety and efficacy of N-Acetyl-L-Leucine (IB1001) for the treatment of Ataxia-Telangiectasia (A-T).

There are two phases to this study: the Parent Study, and the Extension Phase.

The Parent Study evaluates the safety and efficacy of N-Acetyl-L-Leucine (IB1001) for the symptomatic treatment of A-T.

The Extension Phase evaluates the long-term safety and efficacy of IB1001 for the neuroprotective, disease-modifying treatment of A-T.

DETAILED DESCRIPTION:
The primary purpose of the study is to evaluate the safety and efficacy of N-Acetyl-L-Leucine (IB1001) in the treatment of A-T investigating the efficacy in terms of improving symptoms, functioning, and quality of life against the defined endpoints in patients with A-T.

Patients will be assessed during three study phases: a baseline period, a 6-week treatment period, and a 6-week post-treatment washout period. If within 6 weeks prior to the initial screening visit, a patient has received any of the prohibited medications defined in the eligibility criteria (irrespective of the preceding treatment duration) a wash-out study-run in of 6 weeks is required prior to the first baseline assessment.

All patients will receive the study drug during this study.

For each individual patient, the study lasts for approximately 3.5 - 4 months during which there are 6 study visits to the study site.

This Extension Phase allows patients who have completed the Parent Study to, at the discretion of the Principal Investigator (PI), continue treatment with N-Acetyl-L-Leucine (IB1001). Patients will receive treatment with IB1001 for two one-year treatment periods, separated by a 6-week washout. All patients will receive the study drug during the treatment period. For each individual patient, the Extension Phase lasts for approximately 25.5 months, during which there are 6 visits to the study site.

ELIGIBILITY:
Inclusion Criteria

Individuals who meet all of the following criteria are eligible to participate in the study:

1. Written informed consent signed by the patient and/or their legal representative/ parent
2. Male or female aged ≥6 years with a confirmed diagnosis of A-T at the time of signing informed consent.
3. Females of childbearing potential, defined as a premenopausal female capable of becoming pregnant, will be included if they are either sexually inactive (sexually abstinent for 14 days prior to the first dose continuing through 28 days after the last dose) or using one of the following highly effective contraceptives (i.e. results in <1% failure rate when used consistently and correctly) 14 days prior to the first dose continuing through 28 days after the last dose:

   1. intrauterine device (IUD);
   2. surgical sterilization of the partner (vasectomy for 6 months minimum);
   3. combined (estrogen or progestogen containing) hormonal contraception associated with the inhibition of ovulation (either oral, intravaginal, or transdermal);
   4. progestogen-only hormonal contraception associated with the inhibition of ovulation (either oral, injectable, or implantable);
   5. intrauterine hormone-releasing system (IUS);
   6. bilateral tubal occlusion.
4. Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy;

   OR

   be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status. FSH analysis for postmenopausal women will be done at screening. FSH levels should be in the postmenopausal range as determined by the central laboratory.
5. Non-vasectomized male patient agrees to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication and the female partner agrees to comply with inclusion criteria 3 or 4. For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.
6. If male, the patient agrees not to donate sperm from the first dose until 90 days after dosing.
7. Patients must fall within:

   a) A SARA score of 5 ≤ X ≤ 33 points (out of 40) AND i. Within the 2-7 range (out of 0-8 range) of the Gait subtest of the SARA scale OR ii. Be able to perform the 9 Hole Peg Test with Dominant Hand (9HPT-D) (SCAFI subtest) in 20 ≤ X ≤150 seconds.
8. Weight ≥15 kg at screening.
9. Patients are willing to disclose their existing medications/therapies for (the symptoms) of A-T, including those on the prohibited medication list. Non-prohibited medications/therapies (e.g. concomitant speech therapy, and physiotherapy) are permitted provided:

   1. The Investigator does not believe the medication/therapy will interfere with the study protocol/results
   2. Patients have been on a stable dose/duration and type of therapy for at least 6 weeks before Visit 1 (Baseline 1)
   3. Patients are willing to maintain a stable dose/do not change their therapy throughout the duration of the study.
10. An understanding of the implications of study participation, provided in the written patient information and informed consent by patients or their legal representative/parent, and demonstrates a willingness to comply with instructions and attend required study visits (for children this criterion will also be assessed in parents or appointed guardians).

Exclusion Criteria

Individuals who meet any of the following criteria are not eligible to participate in the study:

1. Asymptomatic patients
2. Patient has clinical features of A-T, but a completely negative result on a previous genetic test for A-T.
3. Patients who have any of the following:

   1. Chronic diarrhea;
   2. Unexplained visual loss;
   3. Malignancies;
   4. Insulin-dependent diabetes mellitus.
   5. Known history of hypersensitivity to the N-Acetyl-Leucine (DL-, L-, D-) or derivatives.
   6. History of known hypersensitivity to excipients of Ora-Blend® (namely sucrose, sorbitol, cellulose, carboxymethylcellulose, xanthan gum, carrageenan, dimethicone, methylparaben, and potassium sorbate).
4. Simultaneous participation in another clinical study or participation in any clinical study involving administration of an investigational medicinal product (IMP; 'study drug') within 6 weeks prior to Visit 1.
5. Patients with a physical or psychiatric condition which, at the investigator's discretion, may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the clinical study.
6. Known clinically-significant (at the discretion of the investigator) laboratories in hematology, coagulation, clinical chemistry, or urinalysis, including, but not limited to:

   1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5x upper limit of normal (ULN);
   2. Total bilirubin >1.5x ULN, unless Gilbert's syndrome is present in which case total bilirubin >2x ULN.
7. Known or persistent use, misuse, or dependency of medication, drugs, or alcohol.
8. Current or planned pregnancy or women who are breastfeeding.
9. Patients with severe vision or hearing impairment (that is not corrected by glasses or hearing aids) that, at the investigator's discretion, interferes with their ability to perform study assessments.
10. Patients who have been diagnosed with arthritis or other musculoskeletal disorders affecting joints, muscles, ligaments, and/or nerves that by themselves affects patient's mobility and, at the investigator's discretion, interferes with their ability to perform study assessments.
11. Patients unwilling and/or not able to undergo a 6-week washout period from any of the following prohibited medication prior to Visit 1 (Baseline 1) and remain without prohibited medication through Visit 6.

    1. Aminopyridines (including sustained-release form);
    2. N-Acetyl-DL-Leucine (e.g. Tanganil®);
    3. N-Acetyl-L-Leucine (prohibited if not provided as IMP);
    4. Riluzole;
    5. Gabapentin;
    6. Varenicline;
    7. Chlorzoxazone;
    8. Sulfasalazine;
    9. Rosuvastatin.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Impression of Change in Severity (CI-CS) | CI-CS comparing Baseline (Day 1) with IB1001 verses the end of 6-weeks treatment with IB1001 (Approximately Day 42) MINUS the CI-CS comparing the end of 6-weeks treatment with IB1001 (Approximately Day 42) verses the end of 6-weeks post-treatment washout
  The primary evaluation of the CI-CS will be performed by two independent neurologists whose assessments will be based on videos of the anchor test taken at each visit. These raters will be blinded to the treatment phases and the chronological order of the videos to reduce detection and performance bias.
  The CI-CS assessment will instruct the blinded rater to consider: 'compared to the first video, how has the severity of their performance on the 9HPT-D or 8MWT changed (improved or worsened) in 6-weeks as observed in the second video?'
  The CI-CS is evaluated on a 7 point Likert scale (+3=significantly improved to -3= significantly worse).

SECONDARY OUTCOMES:
Spinocerebellar Ataxia Functional Index (SCAFI) | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The SCAFI scale is a validated ataxia rating scale and is an objective measure of ataxia and physical functioning which consists of three subscales: the 8 Meter Walk Test (8MWT), the 9-hole peg test with both dominant and non-dominant hands (9HPT-D; 9HPT-ND) and the "PATA" test to measure speech performance.
  For the 8MWT and 9HPT tests, a lower score/time indicates a clinical improvement. A higher "PATA" test score indicates improvement in speech performance.
  The SCAFI total score, and three subscales (8MWT, 9HPT-D, and PATA) are reported for statistical analysis.
Change in the Scale for Assessment and Rating of Ataxia (SARA) score | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The SARA scale is an eight-item clinical rating scale (gait, stance, sitting, speech, fine motor function and taxis) with a total score range of 0-40, where 0 is the best neurological status and 40 the worst.
  SARA is a reliable and validated clinical scale with a high internal consistency that measures the severity and progression of ataxia.
EuroQuol- 5 Dimension (EQ-5D) Quality of Life Scale | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The EQ-5D is a standardized measure of health status consists of two parts: a multiple-choice questionnaire (descriptive system) and a visual analogue scale.
  The EQ-5D descriptive system comprises the following 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Investigator's Clinical Global Impressions (CGI) | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The CGI Scale is a widely validated scale that long been implemented in neurodegenerative disease trials to provide an index of clinical importance that cannot be obtained from quantitative assessment measures.
  The CGI comprises of two companion one-item measures evaluating: (A) The severity of the patient's condition and (B) the change from the initiation of treatment. Both measures are evaluated on a 1 to 7 point Likert scale, with 1 indicating the best clinical status and 7 indicating the worst.
Parent/Caregiver's Clinical Global Impressions (CGI) | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The CGI Scale is a widely validated scale that long been implemented in neurodegenerative disease trials to provide an index of clinical importance that cannot be obtained from quantitative assessment measures.
  The CGI comprises of two companion one-item measures evaluating: (A) The severity of the patient's condition and (B) the change from the initiation of treatment. Both measures are evaluated on a 1 to 7 point Likert scale, with 1 indicating the best clinical status and 7 indicating the worst.
Patient's Clinical Global Impressions (CGI) if able | Baseline (Day 1) to end of treatment with IB1001 (Approximately Day 42); End of treatment with IB1001 (Approximately Day 42) to the end of post-treatment washout (Approximately Day 84)
  The CGI Scale is a widely validated scale that long been implemented in neurodegenerative disease trials to provide an index of clinical importance that cannot be obtained from quantitative assessment measures.
  The CGI comprises of two companion one-item measures evaluating: (A) The severity of the patient's condition and (B) the change from the initiation of treatment. Both measures are evaluated on a 1 to 7 point Likert scale, with 1 indicating the best clinical status and 7 indicating the worst.

CONTACTS AND LOCATIONS:
Locations (5):
- University of California - Los Angeles, Los Angeles, California, United States
- Germany (2):
  - University of Giessen, Giessen
  - Ludwig Maximilian University of Munich, München
- Hospital Universitario La Paz, Madrid, Spain, Spain
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brueggemann A, Bicvic A, Goeldlin M, Kalla R, Kerkeni H, Mantokoudis G, Abegg M, Kolnikova M, Mohaupt M, Bremova-Ertl T. Effects of Acetyl-DL-Leucine on Ataxia and Downbeat-Nystagmus in Six Patients With Ataxia Telangiectasia. J Child Neurol. 2022 Jan;37(1):20-27. doi: 10.1177/08830738211028394. Epub 2021 Oct 7. PMID 34620022
- [Derived] Churchill GC, Strupp M, Factor C, Bremova-Ertl T, Factor M, Patterson MC, Platt FM, Galione A. Acetylation turns leucine into a drug by membrane transporter switching. Sci Rep. 2021 Aug 4;11(1):15812. doi: 10.1038/s41598-021-95255-5. PMID 34349180
- [Derived] Fields T, Patterson M, Bremova-Ertl T, Belcher G, Billington I, Churchill GC, Davis W, Evans W, Flint S, Galione A, Granzer U, Greenfield J, Karl R, Kay R, Lewi D, Mathieson T, Meyer T, Pangonis D, Platt FM, Tsang L, Verburg C, Factor M, Strupp M. A master protocol to investigate a novel therapy acetyl-L-leucine for three ultra-rare neurodegenerative diseases: Niemann-Pick type C, the GM2 gangliosidoses, and ataxia telangiectasia. Trials. 2021 Jan 22;22(1):84. doi: 10.1186/s13063-020-05009-3. PMID 33482890